CLINICAL TRIAL: NCT02684123
Title: A Randomized Placebo-controlled Single Center Pilot Study of the Safety and Efficacy of Apremilast in Subjects With Moderate to Severe Alopecia Areata
Brief Title: Pilot Study of the Safety and Efficacy of Apremilast in Subjects With Moderate to Severe Alopecia Areata
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Emma Guttman, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCO 15-1817
Record Dates: First submitted 2016-02-11; First posted 2016-02-17 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Alopecia Areata
Keywords: Alopecia areata
MeSH Terms: conditions — Alopecia Areata | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apremilast (Active Comparator): Apremilast 30mg twice daily
  Interventions: Drug: Apremilast
- Placebo (Placebo Comparator): Placebo pills twice daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apremilast — Subjects will get drug or placebo
  Other Names: Otezla
  Arms: Apremilast
Drug: Placebo
  Arms: Placebo

SUMMARY:
Alopecia areata (AA) is a medical condition, in which the hair falls out in patches. The hair can fall out on the scalp or elsewhere on the face and body.

Alopecia areata is an autoimmune skin disease, which means that the immune system is recognizing the hair follicles as foreign and attacking them, causing round patches of hair loss. It can progress to total scalp hair loss (alopecia totalis) or complete body hair loss (alopecia universalis). The scalp is the most commonly affected area, but the beard or any hair-bearing site can be affected alone or together with the scalp. Alopecia areata occurs in males and females of all ages, and is a highly unpredictable condition that tends to recur. Alopecia areata can cause significant distress to both patients and their families.

In this study, the aim to assess the effects of a new treatment called apremilast in patients with alopecia areata. A total of 30 patients will be included in the study, which will run for a total of 52 weeks.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled pilot study consisting of two phases. A total of 30 subjects with moderate to severe alopecia areata (including universalis and totalis) involving 50-100% of the scalp will be enrolled. A possible maximum of 15 patients (approximately 7 patients each) with current episodes of AA totalis / universalis may be included in this study.

In Phase 1, subjects will be randomized (2:1) to either receive apremilast or placebo for 24 weeks.

In Phase 2, eligible subjects will receive apremilast from Week 24 through Week 48. The following subjects will be eligible to enter into Phase 2:

1. Subjects who received placebo in Phase 1 of the study
2. Subjects who received apremilast in Phase 1 of the study, and who achieved a minimum of 50% regrowth (SALT50) at Week 24, compared to Baseline.

ELIGIBILITY:
Inclusion Criteria:

Males or females, 18 years or older at the time of signing the informed consent document.

Understand and voluntarily sign an informed consent document prior to any study-related assessments/procedures are conducted.

Able to adhere to the study visit schedule and other protocol requirements. Subject with a diagnosis of patchy scalp alopecia areata present for at least 6 months, and up to a maximum of 10 years.

Patients with ≥50% and <95% total scalp hair loss at Baseline as measured using the SALT score to qualify as moderate to severe AA; and 95%-100% scalp hair loss to qualify as AA totalis/universalis.

Must meet the following laboratory criteria White blood cell count ≥ 3000/mm3 (≥ 3.0 x 109/L) and < 14,000/mm3 (< 14 x 109/L). Platelet count ≥ 100,000/μL (≥ 100 x 109/L). Serum creatinine ≤ 1.5 mg/dL (≤ 132.6 μmol/L). AST (SGOT) and ALT (SGPT) ≤ 2 x upper limit of normal (ULN). If the initial test shows ALT or AST > 2 times the ULN, one repeat test is allowed during the Screening Phase.

Total bilirubin ≤ 2 mg/dL (34 μmol/L). If the initial test shows total bilirubin > 2 mg/dL (34 μmol/L), one repeat test is allowed during the Screening Phase.

Hemoglobin ≥ 10 g/dL (≥ 6.2 mmol/L).

Females of childbearing potential (FCBP) must have a negative pregnancy test at Screening and Baseline. While on investigational product and for at least 28 days after taking the last dose of investigational product (IP), FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy;

OR

Option 2: Male or female condom (latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]); plus spermicide PLUS one additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.

Male subjects (including those who have had a vasectomy) who engage in activity in which conception is possible must use barrier contraception (male latex condom or nonlatex condom NOT made out of natural [animal] membrane [for example, polyurethane]) while on IP and for at least 28 days after the last dose of IP.

No evidence of hair regrowth present at Baseline.

EXCLUSION CRITERIA:

The presence of any of the following will exclude a subject from enrollment:

Clinically significant (as determined by the investigator) cardiac, endocrine, pulmonary, neurologic, psychiatric, hepatic, renal, hematologic, or immunologic disease, or other major uncontrolled diseases that will affect the health of the subject during the study or interfere with the interpretation of study results.

Hepatitis B surface antigen positive at Screening (Visit 1). Hepatitis C antibody positive at Screening (Visit 1). History of positive human immunodeficiency virus (HIV), or congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID]). Subjects deemed at risk by the study investigator, may also undergo testing for human immunodeficiency virus (HIV). Subjects deemed at risk include those with a history of injection drug use, homosexual subjects, and subjects with known sexual contact with an HIV positive partner.

Active TB or a history of inadequately treated TB. Active substance abuse or a history of substance abuse within six months prior to Screening.

Pregnant or breast feeding. History of allergy to any component of the IP.

Major surgery within eight weeks prior to Screening (Visit 1) and/or planned surgery during the length of the study.

Malignancy or history of malignancy, except for:

treated (ie, cured) basal cell or squamous cell in situ skin carcinomas; treated (ie, cured) cervical intraepithelial neoplasia (CIN) or carcinoma in situ of the cervix with no evidence of recurrence within 5 years prior to Screening (Visit 1).

Unstable asthma (eg, acute episodes of exacerbation [nocturnal episodes, sudden episodes triggered by unidentifiable factors] despite a stable regimen of anti-asthmatic medications); prior episode(s) of life-threatening asthma; or asthma that requires inhaled budesonide or equivalent at >1200 μg/day or fluticasone propionate at > 880 μg/day along with another anti-asthmatic drug such as a long-acting beta-agonist.

A history of and/or concurrent condition of serious hypersensitivity (eg, anaphylaxis) to drugs, foods, or other allergens without access to emergency rescue medication such as epinephrine.

Persistent or recurring bacterial infection requiring systemic antibiotics, or clinically significant viral or fungal infections, within two weeks of Screening (Visit 1). Any treatment for such infections must have been completed at least two weeks prior to the Screening Visit and no new/recurrent infections should have occurred prior to the Baseline Visit.

Active skin infection requiring systemic antimicrobials at Baseline/Randomization (Visit 2).

Skin lesion(s) due to conditions other than AA that would interfere with the study specified assessments.

Prior treatment with apremilast, or participation in a clinical study involving apremilast.

Use of phototherapy (ie, UVB, UVA) or systemic immunosuppressive drugs (including, but not limited to, cyclosporine, corticosteroids, mycophenolate mofetil, azathioprine, Methotrexate, or tacrolimus), or oral preparations of herbal immunomodulatory medications within four weeks prior to Baseline/Randomization (Visit 2).

Use of interferon-γ within 12 weeks prior to Baseline/Randomization (Visit 2). Use of abatacept, adalimumab, certolizumab pegol, etanercept, golimumab, infliximab, or tocilizumab within 12 weeks prior to Baseline/Randomization (Visit 2).

Use of oral janus kinase (JAK) inhibitors (e.g. tofacitinib, ruxolitinib) within 12 weeks prior to Baseline/Randomization (Visit 2).

Use of omalizumab, rituximab, ustekinumab, alefacept, briakinumab, or other therapeutic antibody products within 24 weeks prior to Baseline/Randomization (Visit 2).

Use of any investigational drug within four weeks or five PK or PD half lives (whichever is longer) prior to Baseline/Randomization (Visit 2).

Use of topical corticosteroid preparations, topical calcineurin inhibitors, or other topical preparations with immunomodulatory properties within 2 weeks prior to Baseline/Randomization (Visit 2).

Prior history of suicide attempt at any time in the subject's lifetime prior to Baseline (Visit 2) or major psychiatric illness requiring hospitalization within 3 years prior to Baseline (Visit 2).

History of male or female pattern hair loss Ludwig stage III or Hamilton > stage V.

Patients in whom the diagnosis of alopecia areata is in question, or subjects with scarring alopecia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-02; Primary Completion 2017-09-15 (Actual); Study Completion 2017-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Guttman, MD, PhD, Principal Investigator — ISMMS
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haider AS, Lowes MA, Suarez-Farinas M, Zaba LC, Cardinale I, Khatcherian A, Novitskaya I, Wittkowski KM, Krueger JG. Identification of cellular pathways of "type 1," Th17 T cells, and TNF- and inducible nitric oxide synthase-producing dendritic cells in autoimmune inflammation through pharmacogenomic study of cyclosporine A in psoriasis. J Immunol. 2008 Feb 1;180(3):1913-20. doi: 10.4049/jimmunol.180.3.1913. PMID 18209089
- [Background] Alkhalifah A. Alopecia areata update. Dermatol Clin. 2013 Jan;31(1):93-108. doi: 10.1016/j.det.2012.08.010. Epub 2012 Oct 2. PMID 23159179
- [Background] Croxford AL, Mair F, Becher B. IL-23: one cytokine in control of autoimmunity. Eur J Immunol. 2012 Sep;42(9):2263-73. doi: 10.1002/eji.201242598. PMID 22949325
- [Background] Vaccaro M, Cannavo SP, Imbesi S, Cristani M, Barbuzza O, Tigano V, Gangemi S. Increased serum levels of interleukin-23 circulating in patients with non-segmental generalized vitiligo. Int J Dermatol. 2015 Jun;54(6):672-4. doi: 10.1111/ijd.12392. Epub 2014 Nov 27. PMID 25427848

RESULTS

PARTICIPANT FLOW:
Groups:
- Apremilast: 30mg twice daily
- Placebo: pills twice daily
Period: Phase 1
Arm/Group | Apremilast | Placebo
Started | 20 | 10
Completed | 12 | 9
Not Completed | 8 | 1
Not completed — Lack of Efficacy | 5 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Period: Eligibility Determination for Phase 2
Arm/Group | Apremilast | Placebo
Started | 12 | 9
Completed | 1 | 9
Not Completed | 11 | 0
Period: Phase 2
Arm/Group | Apremilast | Placebo
Started | 1 | 9
Completed | 0 | 1
Not Completed | 1 | 8
Not completed — Lack of Efficacy | 1 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apremilast | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (14.4) | 44.15 (16.9) | 41.8 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 5 | 21
  Male | 4 | 5 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 17 | 9 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 17 | 9 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Duration of AA [Mean (Standard Deviation); unit: years] | 4.3 (2.7) | 6.6 (2.8) | 5.1 (2.9)
SALT score [Mean (Standard Deviation); unit: units on a scale] — Scalp is divided into 4 areas namely, Vertex - 40% (0.4) of scalp surface area; right profile of scalp - 18% (0.18) of scalp surface area; left profile of scalp - 18% (0.18) of scalp surface area; Posterior aspect of scalp - 24% (0.24) of scalp surface area. Percentage of hair loss in any of these areas is percentage hair loss multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all above mentioned areas.
  units on a scale | 88.0 (19.8) | 87.7 (16.1) | 87.8 (17.1)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With SALT50
Description: Number of patients achieving 50% or greater improvement in their Severity of Alopecia Tool (SALT) score (SALT50) at Week 24
  SALT50 is defined as the percent of patients achieving >=50% reduction in SALT score compared to baseline.
  Scalp is divided into 4 areas namely, Vertex - 40% (0.4) of scalp surface area; right profile of scalp - 18% (0.18) of scalp surface area; left profile of scalp - 18% (0.18) of scalp surface area; Posterior aspect of scalp - 24% (0.24) of scalp surface area. Percentage of hair loss in any of these areas is percentage hair loss multiplied by percent surface area of the scalp in that area. SALT score is the sum of percentage of hair loss in all above mentioned areas.
Time Frame: Baseline and Week 24
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 1 | 9
Participants | 1 | 1

2. Secondary Outcome: Mean Change in SALT Score
Description: Mean percent change in SALT score at 4, 8, 12, 16, 20, and 24 weeks as compared to baseline
Time Frame: Baseline and week 4, 8, 12, 16, 20, 24
Population: Data for participants who returned for particular visits.
Measure: Mean (Standard Error); unit: Mean percent change
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 20 | 10
Mean percent change
  Week 4: number analyzed (Participants) | 18 | 10
  Week 4 | -0.13 (0.56) | -0.11 (0.11)
  Week 8: number analyzed (Participants) | 15 | 9
  Week 8 | -2.39 (2.58) | -2.86 (1.47)
  Week 12: number analyzed (Participants) | 15 | 9
  Week 12 | -0.99 (1.52) | -4.07 (2.21)
  Week 16: number analyzed (Participants) | 14 | 8
  Week 16 | -8.15 (7.37) | -10.55 (6.68)
  Week 20: number analyzed (Participants) | 13 | 8
  Week 20 | 1.17 (2.00) | -9.92 (6.48)
  Week 24: number analyzed (Participants) | 12 | 9
  Week 24 | -1.45 (5.39) | -9.01 (6.37)

3. Secondary Outcome: Phase 2: Number of Patients Achieving aaPGA Score of 3 or Above
Description: Number of subjects achieving an alopecia areata Physician's Global Assessment (aaPGA) score of 3 or above at Weeks 24 (0, no regrowth; 1, <25% of regrowth; 2, 25%-49% of regrowth; 3, 50%-74% of regrowth; 4, 75%-99% of re- growth; 5, 100% of regrowth).
Time Frame: Week 24 and Week 48
Population: Only those who completed treatments as respective week analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 1 | 9
Participants
  week 24 | 1 | 1
  week 48 | 0 | 1

4. Secondary Outcome: Phase 2: Change in AASIS
Description: Change from Baseline in the Alopecia Areata Symptom Impact Scale (AASIS) at Weeks 24 and Week 48 The AASIS is a 13-items disease-specific patient-reported outcomes measure that asks participants about symptoms related to alopecia areata and how these symptoms interfere with daily functioning. Total scale ranges from 0-130, with higher score indicating more symptoms.
Time Frame: Week 24 and Weeks 48
Population: Data for participants who returned for particular visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 19 | 10
score on a scale
  Baseline | 56.79 (30.44) | 51.4 (25.68)
  Week 24: number analyzed (Participants) | 11 | 7
  Week 24 | 48.0 (29.58) | 53.57 (23.59)
  week 48: number analyzed (Participants) | 0 | 3
  week 48 |  | 75.67 (3.79)

5. Secondary Outcome: Phase 2: AA-QoL
Description: Change from baseline in the Alopecia Areata Quality of Life questionnaire (AA-QoL) at Weeks 24 and Weeks 48.
  Total scale from 0 to 100, with higher score indicating better quality of life.
Time Frame: Baseline, Week 24 and Weeks 48
Population: Data for participants who returned for particular visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale
  Baseline | 30.75 (11.88) | 34.0 (20.93)
  Week 24: number analyzed (Participants) | 11 | 7
  Week 24 | 29.55 (11.52) | 27.14 (11.55)
  week 48: number analyzed (Participants) | 0 | 3
  week 48 |  | 35.33 (2.08)

6. Secondary Outcome: Phase 2: Semiquantitative Score
Description: Semiquantitative score using SALT subclasses (0, no hair loss; 1, <25% hair loss; 2, 25%-49% hair loss; 3, 50%-74% hair loss; 4, 75%-99% hair loss; 5, 100% hair loss) at week 24 and week 48 compared to baseline
Time Frame: Baseline, Week 24 and Weeks 48
Population: Data for participants who returned for particular visits
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Apremilast | Placebo
Number analyzed (Participants) | 20 | 10
score on a scale
  Baseline | 4.35 (0.75) | 4.3 (0.82)
  Week 24: number analyzed (Participants) | 12 | 9
  Week 24 | 4.42 (1.16) | 4.1 (1.27)
  week 48: number analyzed (Participants) | 0 | 3
  week 48 |  | 3.67 (2.31)

ADVERSE EVENTS:
Time Frame: 48 weeks
Arm/Group | Apremilast | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/10
Other Adverse Events (participants affected / at risk) | 9/20 | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Apremilast (N=20) | Placebo (N=10)
Nausea (Gastrointestinal disorders) | 4 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 1
Upper respiratory tract infections (Infections and infestations) | 1 | 1
Fatigue (General disorders) | 0 | 1
Tinea pedis (Skin and subcutaneous tissue disorders) | 1 | 0
Diffuse arthralgias (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (General disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 0
Hypertension (Cardiac disorders) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1

LIMITATIONS AND CAVEATS:
This was an exploratory study. Future studies with a larger sample size are needed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/23/NCT02684123/Prot_SAP_000.pdf